CLINICAL TRIAL: NCT03251508
Title: Salvage Peanut Oral Immunotherapy Study: A Single-arm, Open Label Trial of Peanut Flour With 6 Month Active Treatment and 6 Month Follow-up
Brief Title: Salvage Peanut Oral Immunotherapy Study
Acronym: SOIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0195
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2022-12

CONDITIONS: Peanut Allergy
Keywords: Peanut
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peanut OIT/dietary peanut (Experimental): Single arm study with all subjects receiving peanut OIT study drug for the initial 6 months. This is followed by daily ingestion of common dietary foods containing approximately 300 mg of peanut protein for an additional 6 months.
  Interventions: Drug: Peanut OIT

INTERVENTIONS:
Drug: Peanut OIT — Participants will be given increasing doses of the peanut flour as peanut oral immunotherapy (OIT) with increasing doses every 2 weeks over a period of 3 months up to a 300 mg target dose. This 300 mg peanut OIT maintenance dose is then continued daily for 3 months. Participants will then introduce dietary peanut of approximately 300 mg of peanut protein and continue daily ingestion for an additional 6 months.
  Other Names: Peanut flour

SUMMARY:
The purpose of this trial is to study the safety of rescue peanut oral immunotherapy followed by the introduction of dietary peanut for patients with peanut allergy who have lost desensitization during a peanut immunotherapy trial.

DETAILED DESCRIPTION:
Salvage Peanut Oral Immunotherapy Study is a single-arm, open label trial of peanut flour oral immunotherapy (OIT) administered for 6 months followed by introduction of dietary peanut for an additional 6 months.

The peanut OIT phase will involve approximately 3 months of dose escalation up to a maintenance dose of 300 mg peanut protein. This is followed by 3 months of daily maintenance dosing with 300 mg of peanut protein. Patients are then transitioned to the dietary peanut phase ingesting common foods containing approximately 300 mg of peanut protein daily.

Safety will be assessed during both peanut OIT and dietary peanut phases with adverse events recorded including gastrointestinal side effects. They will also be monitored for any anaphylaxis or injectable epinephrine administration. Data regarding compliance with peanut OIT will be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed an immunotherapy trial for peanut allergy within the last 6 months and are unable to tolerate ≥ 300mg of peanut.
* Age 1-65 years of either sex, any race, any ethnicity. Written informed consent from patient or parent/guardian (if < 18 years) with participant's assent.

Exclusion Criteria:

* Current participation in an interventional study for peanut allergy
* History of a severe anaphylactic reaction to peanut, defined as hypoxia, hypotension, or neurologic compromise (cyanosis or SpO2 ≤ 92% at any stage, hypotension, confusion, collapse, loss of consciousness, or incontinence)
* Eosinophilic or other inflammatory (e.g. celiac) gastrointestinal disease
* Severe asthma (2007 NHLBI Criteria Steps 5 or 6 , Appendix 2)
* Use of B blockers (oral), angiotensin-converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARB) or calcium channel blockers
* Significant medical condition (e.g., liver, kidney, gastrointestinal, cardiovascular, hematologic, or pulmonary disease) which would put the subject at risk for induction of severe food reactions.

Pregnancy or lactation.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Kim, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Peanut Oral Immunotherapy/Dietary Peanut: Subjects receiving peanut flour oral immunotherapy (OIT) up to maintenance dose of 300 mg over initial 6 months. This is followed by daily ingestion of common dietary foods containing approximately 300 mg of peanut protein for an additional 6 months.
Period: Peanut Oral Immunotherapy (Months 1-6)
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Started | 15
Completed | 11
Not Completed | 4
Period: Dietary Peanut (Months 7-12)
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label Peanut Oral Immunotherapy/Dietary Peanut: Subjects receiving peanut oral immunotherapy (OIT) up to maintenance dose of 300 mg over initial 6 months. This is followed by daily ingestion of common dietary foods containing approximately 300 mg of peanut protein for an additional 6 months.
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.9 [4.7 to 13.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Prior Immunotherapy Study [Count of Participants; unit: Participants]
  Peanut Oral Immunotherapy (OIT) | 5
  Peanut Sublingual Immunotherapy (SLIT) | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events During the 2-stage Study Sequence (Safety)
Description: Percentage of participants experiencing an adverse event related to peanut oral immunotherapy (OIT) or dietary peanut ingestion
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
percentage of participants | 60

2. Secondary Outcome: Percentage of Missed Doses During the 2-stage Study Sequence (Compliance)
Description: Evaluation of patient compliance with a 2-stage peanut oral immunotherapy (OIT) and dietary peanut protocol as measured by the percentage of doses missed over the entire 2-stage study protocol sequence.
Time Frame: 12 months
Measure: Number; unit: percentage of missed doses
Units Other Than Participants: immunotherapy & dietary peanut doses
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
Number analyzed (immunotherapy & dietary peanut doses) | 5103
percentage of missed doses | 1.2

3. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events During the Peanut Oral Immunotherapy Stage
Description: Evaluation of peanut oral immunotherapy (OIT) safety measured by the percentage of participants experiencing an adverse event related to peanut OIT during the peanut oral immunotherapy (OIT) stage of the 2-stage Peanut Oral Immunotherapy/Dietary Peanut protocol.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
percentage of participants | 60

4. Secondary Outcome: Percentage of Missed Doses During the Peanut Oral Immunotherapy Stage
Description: Evaluation of patient compliance measured by the percentage of doses missed during the peanut oral immunotherapy (OIT) stage of the 2-stage Peanut Oral Immunotherapy/Dietary Peanut protocol.
Time Frame: 6 months
Measure: Number; unit: percentage of missed doses
Units Other Than Participants: oral immunotherapy doses
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
Number analyzed (oral immunotherapy doses) | 2863
percentage of missed doses | 2.1

5. Secondary Outcome: Percentage of Participants Utilizing Emergency Epinephrine Use During the 2-Stage Study Sequence (Safety)
Description: Percentage of participants utilizing epinephrine for treatment of an adverse event related to peanut oral immunotherapy (OIT) or dietary peanut
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
percentage of participants | 0

6. Secondary Outcome: Percentage of Participants Experiencing Gastrointestinal Adverse Events During the 2-stage Study Sequence (Safety)
Description: Percentage of participants experiencing a gastrointestinal adverse event related to peanut oral immunotherapy (OIT) or dietary peanut
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
percentage of participants | 53.33

7. Secondary Outcome: Percentage of Participants Withdrawing During the 2-stage Study Sequence Due to Gastrointestinal Adverse Events (Safety)
Description: Percentage of participants withdrawing from the study due to a gastrointestinal adverse event related to peanut oral immunotherapy (OIT) or dietary peanut
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Open-label Peanut Oral Immunotherapy/Dietary Peanut
Number analyzed (Participants) | 15
percentage of participants | 13.33

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of signing consent through the completion of 12 month treatment protocol.
Description: Dose escalation symptoms were recorded by study coordinators. Home OIT and dietary peanut symptoms were reported by parents through home diaries.
Groups:
- Open-label Peanut OIT/Dietary Peanut: Subjects receiving peanut OIT up to maintenance dose of 300 mg over initial 6 months. This is followed by daily ingestion of common dietary foods containing approximately 300 mg of peanut protein for an additional 6 months.
Arm/Group | Open-label Peanut OIT/Dietary Peanut
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 9/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Peanut OIT/Dietary Peanut (N=15)
Skin adverse events (Skin and subcutaneous tissue disorders) | 5
Upper respiratory adverse events (Respiratory, thoracic and mediastinal disorders) | 3
Lower respiratory adverse events (Respiratory, thoracic and mediastinal disorders) | 2
Gastrointestinal adverse events (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03251508/Prot_SAP_000.pdf